CLINICAL TRIAL: NCT05146193
Title: AI-Powered Scoliosis Auto-Analysis System Multicenter Development and Validations
Status: Recruiting | Type: Observational
Sponsor: The University of Hong Kong (Other)
Collaborators: Peking Union Medical College (Other); Peking University Third Hospital (Other); Beijing Chao Yang Hospital (Other); University of Malaya (Other); Nara Medical University (Other); Hamamatsu University (Other); Ruijin Hospital (Other); Huashan Hospital (Other); Zhejiang University (Other); Ji Shui Tan Hospital (Unknown)
Responsible Party: Principal Investigator, Dr. Jason Pui Yin Cheung, Clinical Associate Professor, The University of Hong Kong
Other Study IDs: AI_Scoliosis
Record Dates: First submitted 2021-11-12; First posted 2021-12-06 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Spinal Deformity
Keywords: Adult deformity, scoliosis, spondylolisthesis
MeSH Terms: conditions — Congenital Abnormalities; Scoliosis; Spondylolisthesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- All subjects are diagnosed of having a spinal deformity: Routine care of patients with spinal deformities
  Interventions: Other: Nude back photo

INTERVENTIONS:
Other: Nude back photo — Nude back photo at baseline and at follow-ups for each patient and visual severity and curve type classifications

SUMMARY:
The investigators aim to use artificial intelligence (AI) to help clinicians in diagnosing and assessing spinal deformities.

DETAILED DESCRIPTION:
Background Spinal deformity is a prevalent spinal disorder in both paediatric and adult populations. The spine alignment need to be quantitively assessed for further treatment planning. However, the current practice requires spine surgeons to manually place landmarks of endplates and key vertebrae. The process is laborious and prone to inter- and intra-rater variance. Thus, the investigators have developed an AI-powered spine alignment assessment system (AlignProCARE) to facilitate clinicians in fast, accurate and consistent analytical results.

The investigators aim to test and improve the performance of the spine alignment auto-analysis in all patients with spinal deformities in multiple centers including Malaysia, China, and Japan

Objectives:

1. prospectively test the alignment assessment of patients' spinal deformities with whole spine X-rays (both PA and lateral) and nude back image with the assessment via AlignProCARE.
2. Collect 500 labeled deformity radiographs and nude back images in both PA and lateral views per center. 150 patients need to be followed up with radiographs and nude back photos collected (all parameters measured again).
3. Use transfer learning to update the current AlignProCARE for scoliosis analysis to form AlignProCARE+.

4 Qualitatively analyse the AlignProCARE+ using an independent dataset.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic scoliosis, adult deformity (spondylolisthesis, idiopathic kyphosis, kyphoscoliosis, lordoscoliosis)

Exclusion Criteria:

* Refusal for imaging, postoperative patients

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All subjects with spinal deformities
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2029-02-01 (Estimated); Study Completion 2030-02-01 (Estimated)

PRIMARY OUTCOMES:
Cobb angle | 1 year
  Coronal Cobb angle of the spinal deformity. The most tilted end vertebrae away from the apex will be used for measurement of the Cobb angle.The anteroposterior radiograph is used to assess

SECONDARY OUTCOMES:
Thoracic kyphosis | 1 year
  Thoracic kyphosis T5-12: angle between upper endplate of T5 to lower endplate of T12 in the lateral radiograph
Lumbar lordosis | 1 year
  Lumbar lordosis L1-S1: angle between upper endplate of L1 to top of S1 in the lateral radiograph
Pelvic tilt | 1 year
  Pelvic tilt angle measurement in degrees in the lateral radiograph
Sacral slope | 1 year
  Sacral slope angle measurement in degrees in the lateral radiograph
Pelvic incidence | 1 year
  Pelvic incidence angle measurement in degrees in the lateral radiograph
Maximum thoracic kyphosis | 1 year
  Maximum thoracic kyphosis: angle measurement from the upper endplate of most tilted upper end vertebra to the lower endplate of the lower end vertebra of the thoracic spine in the sagittal plane radiograph
Curve severity | 1 year
  Severity classifications: normal-mild; moderate and severe

CONTACTS AND LOCATIONS:
Overall Officials: Jason Pui Yin Cheung, MD, MS, Principal Investigator — Queen Mary Hospital, Duchess of Kent Children's Hospital
Locations (1):
- Duchess of Kent Children's Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No